CLINICAL TRIAL: NCT02178709
Title: A Phase II Study of Neoadjuvant FOLFIRINOX in Patients With Resectable Pancreatic Ductal Adenocarcinoma With Tissue Collection
Brief Title: A Phase II Study of Neoadjuvant FOLFIRINOX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Anita Turk, Assistant Professor of Clinical Medicine, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUCRO-0473
Record Dates: First submitted 2014-06-24; First posted 2014-07-01 (Estimated); Results first posted 2020-01-31 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-01

CONDITIONS: Resectable Pancreatic Ductal Adenocarcinoma
Keywords: Pancreatic; Cancer; Resectable
MeSH Terms: conditions — Neoplasms | interventions — folfirinox; Oxaliplatin; Leucovorin; Irinotecan; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FOLFIRINOX (Experimental): FOLFIRINOX consists of the following combination of drugs:
  1. Oxaliplatin, 85 mg/m2, IV over 2 hours prior to irinotecan, administered on days 1 and 15 of each 28 day cycle
  2. Leucovorin, 400 mg/m2, IV over 2 hours with irinotecan, administered on days 1 and 15 of each 28 day cycle
  3. Irinotecan, 180 mg/m2, IV over 90 minutes with leucovorin, administered on days 1 and 15 of each 28 day cycle
  4. 5 FU, 400 mg/m2, IV bolus over 2 minutes after irinotecan, administered on days 1 and 15 of each 28 day cycle.
  5. 5FU, 2400 mg/m2, IV infusion over 46 hours after 5FU bolus injection, administered on days 1 and 15 of each 28 day cycle.
  Interventions: Drug: FOLFIRINOX

INTERVENTIONS:
Drug: FOLFIRINOX — FOLFIRINOX consists of the following combination of drugs:
  1. Oxaliplatin, 85 mg/m2, IV over 2 hours prior to irinotecan, administered on days 1 and 15 of each 28 day cycle
  2. Leucovorin, 400 mg/m2, IV over 2 hours with irinotecan, administered on days 1 and 15 of each 28 day cycle
  3. Irinotecan, 180 mg/m2, IV over 90 minutes with leucovorin, administered on days 1 and 15 of each 28 day cycle 4.5 FU, 400 mg/m2, IV bolus over 2 minutes after irinotecan, administered on days 1 and 15 of each 28 day cycle.
  5.5FU, 2400 mg/m2, IV infusion over 46 hours after 5FU bolus injection, administered on days 1 and 15 of each 28 day cycle.
  Other Names: Oxaliplatin (Eloxatin); Leucovorin; Irinotecan (Camptosar); 5 FU (Adrucil)

SUMMARY:
The primary objective of this study is to evaluate the rate of pathologic complete response to neoadjuvant FOLFIRINOX in patients with resectable pancreatic cancer using a tissue collection component.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old at the time of informed consent
2. Able to provide written informed consent and HIPAA authorization
3. ECOG performance status of 0 or 1
4. Patient must be eligible for abdominal surgery
5. Histologically confirmed adenocarcinoma of the pancreas that has been documented to be resectable by standardized radiographic criteria by a pancreatic surgeon
6. Patients must to have tumor tissue collected prior to enrolling on this trial. Up to 10 patients will be accepted with no pre-treatment research tissue collection or tissue collection from an outside institution.

   a.If the tissue is from an outside institution, it must be reviewed at Indiana University Health Pathology Department if a biopsy was performed outside of this institution.
7. Women of childbearing potential definition (WOCBP) must have a negative serum or urine pregnancy test performed within 14 days prior to initiation of FOLFIRINOX.

   Any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) is classified as WOCBP if she meets the following criteria:
   1. Has not undergone a hysterectomy or bilateral oophorectomy; or
   2. Has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
8. WOCBP and men must agree to use adequate contraception prior, to study entry, for the duration of study participation, and 8 weeks after the end of treatment.
9. Patients must have adequate organ function as defined by the following laboratory values at study entry:

   1. Hemoglobin ≥ 9 g/dL (transfusions are acceptable)
   2. ANC ≥ 1.5 x 109/L
   3. Platelets ≥ 100 x 109/L
   4. Creatinine ≤ 1.5 x ULN, or creatinine clearance ≥ 50 mL/min (estimated by Cockcroft-Gault or measured)
   5. Total bilirubin ≤ 1.5 x ULN
   6. AST/ALT ≤ 3 x ULN

Exclusion Criteria:

1. Prior therapy for pancreatic adenocarcinoma
2. Other malignancies within the past 3 years except for the following: adequately treated cervical or vulvar carcinoma in situ, treated basal cell or squamous carcinoma of the skin, superficial bladder tumors (Ta, Tis & T1), ductal carcinoma in situ (DCIS) of the breast and low grade prostate cancer. Any cancer curatively treated >3 years prior to entry with no clinical evidence of recurrence is permitted.
3. Hypersensitivity to 5FU, oxaliplatin (or other platinum agents), irinotecan (or to their excipients).
4. Participation in any investigational drug study within 4 weeks preceding the start of study treatment. Patients are not permitted to participate in another investigational drug study while being treated on this protocol.
5. Inability to receive a port or PICC line.
6. History of or suspected Gilbert's Disease (testing not required if presence is not suspected).
7. Baseline peripheral neuropathy/paresthesia grade ≥ 1.
8. Active hepatitis B, unless patient has been on antiviral agents for at least 2 months (baseline testing not required).
9. Active clinically serious infections (> grade 2).
10. Major surgery or significant traumatic injury within 8 weeks of first study drug. A core pancreatic or liver biopsy does not preclude the patient from the study.
11. Unable or unwilling to discontinue use of ketoconazole or St John's wort. Use of phenytoin, carbamazepine, phenobarbital, rifampin and rifabutin is discouraged, but not contraindicated. If patients require phenytoin, carbamazepine or phenobarbital monitoring of drug levels is suggested during the study.
12. Pregnant or lactating women.
13. Psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-06-03 (Actual); Primary Completion 2018-02-14 (Actual); Study Completion 2019-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael House, M.D., Principal Investigator — Indiana University
Locations (1):
- Indiana University Simon Cancer Center, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FOLFIRINOX
Started | 48
Completed | 32
Not Completed | 16
Not completed — Adverse Event | 5
Not completed — Death | 2
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 2
Not completed — Disease Progression | 5

BASELINE CHARACTERISTICS:
Arm/Group | FOLFIRINOX
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (9.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 43
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Pathologic Complete Response
Description: Pathologic complete response was evaluated using MRI or CT and Evan's criteria for pathologic response following neoadjuvant therapy:
  I: <10% to no tumor cells destroyed IIa: 10-50% of tumor cells destroyed IIb: 50-90% of tumor cells destroyed III: >90% of tumor cells destroyed IIIM: sizable pools of cellular mucin IV: No viable tumor cells (complete pathologic response) IVM: Acellular pools of mucin
Time Frame: Up to 4 months
Population: All patients who received at least two doses of FOLFIRINOX (unless treatment-related toxicity precluded additional doses) and had at least one post-baseline assessment or died before any evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FOLFIRINOX
Number analyzed (Participants) | 43
percentage of participants | 0 [0 to 0]

2. Secondary Outcome: Number of Patients With Treatment-Related Adverse Events Grade 3 or Above
Description: Number of unique patients who had a treatment-related (possible, probable, or definite) adverse event with grade 3 or greater using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: Every 15 days for approximately 6 months
Population: All patients who received at least one dose of FOLFIRINOX.
Measure: Count of Participants; unit: Participants
Arm/Group | FOLFIRINOX
Number analyzed (Participants) | 48
Participants | 14

3. Secondary Outcome: Percentage of Patients Who Successfully Underwent Surgery After Neoadjuvant FOLFIRINOX
Description: The percentage of patients who successfully underwent surgery after neoadjuvant FOLFIRINOX and its 95% confidence interval will be provided.
Time Frame: Up to 4 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FOLFIRINOX
Number analyzed (Participants) | 43
percentage of participants | 76.7 [64.1 to 89.4]

4. Secondary Outcome: Rate of R0 Resection
Description: The percentage of patients with a final margin status of R0 after resection of their primary tumor and its 95% confidence interval will be provided. R0 resection indicates a microscopically margin-negative resection, in which no cancer cells seen microscopically at the primary tumor site.
Time Frame: Up to 4 months
Population: All patients who completed surgery.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FOLFIRINOX
Number analyzed (Participants) | 33
percentage of participants | 75.8 [61.1 to 90.4]

5. Secondary Outcome: Disease Free Survival
Description: Disease free survival is defined as the time from on study date to evidence of tumor recurrence or death from any cause. Patients who remained alive and disease free were censored at their date of last disease evaluation.
Time Frame: Up to 3 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FOLFIRINOX
Number analyzed (Participants) | 43
months | 8.6 [5.1 to 13.4]

6. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from on study date to death due to any cause. Patients who remained alive were censored at their last known alive date. The Kaplan-Meier method was used to determine the median and 95% confidence interval.
Time Frame: Up to 4 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FOLFIRINOX
Number analyzed (Participants) | 43
months | 15.7 [9.1 to 21.7]

7. Secondary Outcome: Objective Response Rate (Percentage of Patients With Complete Response or Partial Response)
Description: Measured by RECIST v1.1 Complete response: Disappearance of all target lesions Partial response: At least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter
  The percentage of patients with objective response and its 95% confidence interval will be provided.
Time Frame: Up to 4 months
Population: Patients who received four treatments of FOLFIRINOX and had at least one post-baseline assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FOLFIRINOX
Number analyzed (Participants) | 34
percentage of participants | 17.7 [4.8 to 30.5]

8. Secondary Outcome: Disease Control Rate (Percentage of Patients With Complete Response, Partial Response, or Stable Disease)
Description: Measured by RECIST v1.1
  Complete response: Disappearance of all target lesions Partial response: At least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter Stable disease: Neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum longest diameter since the treatment started
  The percentage of patients with objective response and its 95% confidence interval will be provided.
Time Frame: Up to 4 months
Population: Patients who received four treatments of FOLFIRINOX and had at least one post-baseline assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FOLFIRINOX
Number analyzed (Participants) | 34
percentage of participants | 88.2 [77.4 to 99.1]

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | FOLFIRINOX
All-Cause Mortality (participants affected / at risk) | 35/48
Serious Adverse Events (participants affected / at risk) | 15/48
Other Adverse Events (participants affected / at risk) | 42/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFIRINOX (N=48)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (4)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (5)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (6)
Death NOS (General disorders) | 2 (2)
Fever (General disorders) | 3 (4)
Sepsis (Infections and infestations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOLFIRINOX (N=48)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Bloating (Gastrointestinal disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 23 (35)
Mucositis oral (Gastrointestinal disorders) | 5 (6)
Nausea (Gastrointestinal disorders) | 21 (29)
Vomiting (Gastrointestinal disorders) | 10 (11)
Fatigue (General disorders) | 29 (41)
Fever (General disorders) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 10 (11)
Hypokalemia (Metabolism and nutrition disorders) | 9 (10)
Dysgeusia (Nervous system disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 16 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-02): https://cdn.clinicaltrials.gov/large-docs/09/NCT02178709/Prot_SAP_000.pdf